CLINICAL TRIAL: NCT05156892
Title: A Phase I/II Trial Investigating the Tolerability, Toxicity and Efficacy of Tamoxifen and SUBA-Itraconazole in Patients With Platinum Resistant Recurrent Epithelial Ovarian Cancer
Brief Title: Tamoxifen and SUBA-Itraconzole Combination Testing in Ovarian Cancer
Acronym: TICTOC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Anthony Joshua, FRACP (Other)
Collaborators: Royal Prince Alfred Hospital, Sydney, Australia (Other); Concord Hospital (Other); Prince of Wales Hospital, Sydney (Other Government); St Vincent's Hospital, Sydney (Other)
Responsible Party: Sponsor-Investigator, Anthony Joshua, FRACP, Head of Medical Oncology, St Vincent's Hospital, Sydney
Organization: St Vincent's Hospital, Sydney (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TICTOC
Record Dates: First submitted 2021-10-19; First posted 2021-12-14 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer; Tamoxifen; SUBA-Itraconazole; Platinum resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Intervention Model Description: Dose Escalation (3+3) design with Dose Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation/ expansion (Experimental): SUBA-itraconazole (oral 150mg twice daily) and escalating dose of Tamoxifen (oral once daily) then expansion cohort
  Interventions: Drug: SUBA-itraconazole; Drug: Tamoxifen

INTERVENTIONS:
Drug: SUBA-itraconazole — 150 mg BD
Drug: Tamoxifen — Dose Escalation:
  Cohort 1: 20 mg OD Cohort 2: 40 mg OD Cohort 3: 60 mg OD
  Dose-Expansion: Recommended dose from dose-escalation phase of study

SUMMARY:
The study's purpose is to understand the effects of a new treatment (suba-itraconazole and tamoxifen) in epithelial ovarian cancer.

Who is it for? Patients may be eligible to join this study with ovarian cancer resistant to platinum-based chemotherapy agents

Study Details:

Participants will receive different doses of tamoxifen and suba-itraconazole to determine the optimal combination dose.

Participants will be seen by the investigators once a week for the first 3 weeks and then once every 4 weeks. Participant will be reviewed by a clinician and undergo regular blood tests, cardiac monitoring and imaging assessments.

DETAILED DESCRIPTION:
A phase 1/2 study of Suba-itraconazole and Tamoxifen in platinum resistant ovarian carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological-based diagnosis of high grade and low grade epithelial ovarian cancer. Patients with clear cell ovarian cancers are not eligible to participate in this study due to higher risk of thromboemboli which could be increased by Tamoxifen.
2. Platinum resistant ovarian cancer with no more than 4 lines of previous systemic therapy (re-treatment with a previous regimen is only counted as 1 line of therapy).
3. Age > 18 years.
4. Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
5. Eastern Cooperative Oncology Group Performance Status of 0 or 1
6. Adequate hematologic and organ function within 14 days before the first study treatment on Day 1 of Cycle 1, defined by the following:

   * Neutrophils (absolute neutrophil count ANC >1.5X10^9/L,)
   * Hemoglobin >9 g/dL
   * Platelet count >100,000/L
   * Serum albumin >3 g/dL
   * Total bilirubin 1.5 ≤the upper limit of normal (ULN) and AST and ALT ≤2.5 XULN, with the following exception:

     * Patients with known Gilbert syndrome who have serum bilirubin ≤3XULN may be enrolled.
     * Patients with documented liver metastasis may have AST and ALT ≤5XULN
   * PTT (or aPTT) and INR ≤1.5XULN (except for patients receiving anticoagulation therapy)
   * Serum creatinine ≤ 1.5XULN or creatinine clearance >50 mL/min based on Cockcroft-Gault glomerular filtration rate estimation: (140 - age) X(weight in kg) X0.85 (if female) 72 X(serum creatinine in mg/dL)
7. Life expectancy of at least 3 months
8. Have at least 1 measurable lesion assessable using standard techniques by RECIST v1.1. Patients without any measurable disease may be enrolled on a case-by-case basis in discussion with study principle investigator
9. At least 4 weeks washout period from previous line of treatment (including hormonal treatment) , 2 weeks from radiotherapy
10. Ability to swallow and retain oral medications (without crushing, dissolving or chewing tablets)
11. Willing and able to comply with all study requirements, including treatment (e.g. able to swallow tablets), timing and/or nature of required assessments

Exclusion Criteria:

1. Patients with any other prior malignancy from which the patient has been disease free for less than 3 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of any site or any other cancer as approved by study principle investigator
2. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic or asymptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
3. History of or current evidence of HIV infection, Viral hepatitis (e.g., positive for hepatitis B surface antigen [HBsAg] or hepatitis C virus [HCV] antibody at screening)
4. Patients with symptomatic central nervous system (CNS) metastasis and/or carcinomatous meningitis. Patients with treated CNS metastases are eligible for this study if not receiving corticosteroids and/or anticonvulsants for at least 7 days prior to first dose of study treatment, and the disease is asymptomatic and radiographically stable for at least 2 weeks after completion of CNS-directed therapy. Patients with untreated stable or asymptomatic brain metastases may be enrolled on a case-by-case basis in discussion with study principal investigator.
5. Patients with existing or past history of deep venous thromboembolism are excluded, unless stable on anticoagulation.
6. Patients with Khorana score of greater than or equal to 3 (see https://www.mdcalc.com/khorana-risk-score-venousthromboembolism- cancer-patients)
7. Known hypersensitivity or contraindication to any component of the study treatment.
8. Inability to comply with study and follow-up procedures.
9. Patients who have not recovered (≤ grade 2) from adverse events related to previous treatments, unless approved by study principle investigator
10. Patients unable to swallow orally administered medications and patients with gastrointestinal impairment that could affect the ability to take or absorption of oral medications including sub-acute or complete bowel obstruction.
11. Participants with uncontrolled intercurrent illness
12. Participants not recovered from all toxicities related to prior anticancer therapies to CTCAE grade<1 apart from alopecia
13. Patients with psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It is a female only study population as it is investigating Ovarian Cancer
Enrollment: 44 (Estimated)
Dates: Start 2022-09-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose of Tamoxifen in combination with Suba-itraconazole | 1 years

SECONDARY OUTCOMES:
To determine overall response rate as determined by RECIST V1.1 and GCIG CA125 response criteria | 2 years
  ORR
To determine the duration of response | 2 years
  DOR
Incidence of Treatment-Emergent Adverse Events via CTCAE v5.0 | 2 years
  Safety
Serum concentration of tamoxifen and derivatives | 2 years
  Cmax
Serum concentration of tamoxifen and derivatives | 2 years
  AUC
Tissue concentration of tamoxifen and derivatives | 2 years
  mg/g
Serum concentration of itraconazole | 2 years
  Cmax
Serum concentration of itraconazole | 2 years
  AUC
Tissue concentration of itraconazole | 2 years
  mg/g

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, FRACP, MBBS, PhD, Principal Investigator — St Vincent's Hospital, Sydney
Locations (1):
- Kinghorn Cancer Centre, St. Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
No Plan to share participant data with individuals outside this trial